CLINICAL TRIAL: NCT02130414
Title: A Multiple Dose, Multi-stage Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Colon Tissue Distribution of Cyclosporine Capsules (CyCol®) Compared to Intravenous Cyclosporine in Healthy Male Volunteers
Brief Title: PK, Safety & Tolerability of CyCol® Versus Sandimmune® in Healthy Subjects
Acronym: CYC102
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sigmoid Pharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CYC102
Record Dates: First submitted 2014-04-22; First posted 2014-05-05 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-05

CONDITIONS: Healthy
Keywords: Cyclosporine; Healthy Volunteers; Immunosuppressive Agents; CyCol; Pharmacokinetics
MeSH Terms: interventions — Cyclosporine; Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Sandimmun® IV (Active Comparator): Sandimmun® IV 2mg/kg as a 24 hour infusion (2mg/kg/day)
  Interventions: Drug: Sandimmun® IV
- CyCol® capsules (Experimental): CyCol®: 75 mg OD & BID for 7 days
  Interventions: Drug: CyCol® capsules
- CyCol® capsules 37.5 mg (Experimental): CyCol®: 37.5 mg OD or BID for 7 days
  Interventions: Drug: CyCol® capsules
- CyCol® capsules, 150 mg (Experimental): CyCol®: 150 mg OD or BID for 7 days
  Interventions: Drug: CyCol® capsules

INTERVENTIONS:
Drug: Sandimmun® IV — 2 mg/kg IV
  Other Names: Cyclosporine A; Sandimmun® concentrate for solution for Infusion
  Arms: Sandimmun® IV
Drug: CyCol® capsules — 37.5 mg CyCol® capsules
  Other Names: Cyclosporine A; oral cyclosporine
  Arms: CyCol® capsules; CyCol® capsules 37.5 mg; CyCol® capsules, 150 mg

SUMMARY:
The aim of this Phase I, single centre, multi stage study is to evaluate the safety, tolerability, pharmacokinetics and relative colonic mucosal concentrations of cyclosporine capsules (CyCol®) compared to intravenous cyclosporine in healthy male volunteers.

DETAILED DESCRIPTION:
This is an open label, multiple-dose, multi-stage pharmacokinetic (PK) study. A maximum of 40 healthy adult male volunteers aged between 18 and 55 years will be enrolled at a single clinical research unit.

For each CyCol® group dosing will last 7 days, whilst the Sandimmun® IV group will have a single dose over 24 hours.

Single dose pharmacokinetics of different doses of CyCol® will be compared to IV Sandimmun®. In addition colonic tissue concentrations will be compared after multiple doses of CyCol® to a single IV dose of Sandimmun®. Concentrations of unchanged cyclosporine and it's metabolites in the faeces will also be explored.

Stage 1 of the study will investigate the 75mg dose (OD and BID) of CyCol® and IV Sandimmun®. Then dependent on results Stages 2 and 3 will investigate either lower (37.5mg) or higher (150mg) dose levels. The dosing regimens chosen for Stages 2 and 3 will be based upon safety and tolerability, systemic exposure and colonic mucosa tissue concentrations observed at other doses.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers, between the ages of 18 and 55 years, inclusive.
* Mass Index (BMI) of 18.5 to 30.0 kg/m2, inclusive; and a total body weight >50 kg (110 lbs).
* Subjects capable of providing written consent.
* Subjects willing to use acceptable method of contraception starting from the first dose and continuing for at least 3 months after the last dose of study drug.
* Subjects who are willing and able to comply with scheduled visits, dosing plan, laboratory tests, and other study procedures.
* Subjects must have a regular bowel movement

Exclusion Criteria:

* Any condition possibly affecting drug absorption (eg, gastrectomy).
* A positive urine drug screen.
* History of significant drug abuse
* History of regular alcohol consumption
* Treatment with an investigational drug within 90 days prior to first dose of study medication.
* If considered clinically significant by the Investigator, screening supine blood pressure 140 mm Hg (systolic) or 90 mm Hg (diastolic), on a single measurement (confirmed by a single repeat, if necessary) following at least 5 minutes of rest.
* 12-lead ECG demonstrating QTcF interval >450 msec or a QRS interval >120 msec at Screening.
* Use of medications :

  * prescription medications (oral and topical) within 14 days prior to first dosing.
  * over-the-counter products including herbal and food supplements within 7 days prior to first dose of study medication
  * injection or implant of any drug within 3 months prior to first dose of study medication
* Use of any drugs known to induce or inhibit hepatic drug metabolism within 30 days prior to administration of the study medication.
* Plasma donation within 7 days prior to dosing.
* History of sensitivity to cyclosporine or other related drugs.
* Subjects with evidence of ongoing (active or carrier status) hepatitis B or C, or human immunodeficiency virus (HIV) infection upon serological testing.
* History of latent or active tuberculosis or exposure to endemic areas within 8 weeks prior to Quantiferon test performed at screening.
* Positive Quantiferon test result
* Subjects who have received or are planning to receive any live virus vaccination within 28 days prior to the first dose of study medication, or planning to receive a vaccination during the course of the study.
* Any evidence of active infection or febrile illness within 7 days of the first dose of study medication
* Presence of fever (body temperature >37.6oC) within 2 weeks prior to first dose of study medication.
* Subjects who are unwilling to refrain from consumption of grapefruit or products containing grapefruit juice or grapefruit-related citrus fruits (eg, starfruit, pomelos) from 7 days prior to the first dose of study medication until completion of all study procedures.
* Unwilling or unable to comply with the guidelines described in this protocol, or a reason which, in the opinion of the Investigator, would prevent the subject from participating in the study.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2014-07; Primary Completion 2015-01 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic variables for cyclosporine (in whole blood) | Day 1 and Day 7
  Area under the concentration-time curve (AUC) from;
  * time zero to the last non-zero concentration (AUC 0-t),
  * time zero extrapolated to infinity (AUC 0-inf),
  * maximum observed concentration (Cmax)
Concentrations (ng/g) of cyclosporine and its metabolites (AM1, AM9, AM4N) in colonic mucosa | Day 2 or Day 7
  Concentrations (ng/g) of cyclosporine and its metabolites (AM1, AM9, AM4N)in colonic mucosal tissue

SECONDARY OUTCOMES:
Safety and Tolerability of CyCol | Day 1 to Day 7
  Percentage of subjects with clinically significant abnormal results

OTHER OUTCOMES:
Amount of unchanged cyclosporine and its metabolites excreted in faeces | Day 1 through Day 7
  To evaluate the amount (ng/g) of unchanged cyclosporine and its metabolites (AM1, AM9, AM4N) excreted in the faeces.

CONTACTS AND LOCATIONS:
Overall Officials: Sigmoid Pharma, Study Director — Sigmoid Pharma